CLINICAL TRIAL: NCT02132351
Title: Acceptability, Reliability and Applicability of Liver Biopsy and Noninvasive Methods for Assessment of Hepatic Fibrosis and Cirrhosis Among Hepatologists; a Web Based Survey
Brief Title: Hepatic Fibrosis Non-invasive Methods Questionnaire
Status: Completed | Type: Observational
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohamed Alboraie, Post graduate researcher, Al-Azhar University
Other Study IDs: MB-1; AlazharU-MB-1 (Other: AlazharU-MB)
Record Dates: First submitted 2014-05-05; First posted 2014-05-07 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-04

CONDITIONS: Cirrhosis; Fibrosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hepatologists: Doctors working as hepatologists

SUMMARY:
Due to the limitations and the invasive nature of liver biopsy, there has been extensive interest in developing non-invasive tests to measure liver fibrosis (1). These are alternatives to liver biopsy that can be used in clinical practice, with benefits in terms of cost, risk, and patient convenience (2). Clinically applicable non-invasive tests include radiological studies, transient elastography (TE), and serum markers. We aim at studying acceptability, reliability, applicability and practical aspects of invasive and noninvasive methods for assessment of hepatic fibrosis and cirrhosis among hepatologists.

DETAILED DESCRIPTION:
Due to the limitations and the invasive nature of liver biopsy, there has been extensive interest in developing non-invasive tests to measure liver fibrosis (1). These are alternatives to liver biopsy that can be used in clinical practice, with benefits in terms of cost, risk, and patient convenience (2). Clinically applicable non-invasive tests include radiological studies, transient elastography (TE), and serum markers. We aim at studying acceptability, reliability, applicability and practical aspects of invasive and noninvasive methods for assessment of hepatic fibrosis and cirrhosis among hepatologists.

Methods:

The study is a survey study among hepatologists. Four thousand hepatologists will be invited to participate in the questionnaire through e-mail invitations to answer 50 questions of the questionnaire. The questionnaire will be hosted on Survey monkey website and results will be analyzed to get the consensus opinion of participants for the use of invasive and non-invasive methods for assessment of hepatic fibrosis and cirrhosis and factors affecting their preferences.

Statistical analysis plan Analysis of data will be performed using Statistical Package for Scientific Studies 17 for Windows. Description of qualitative variables will be in the form of numbers (No.) and percent (%). Description of quantitative variables will be in the form of mean, standard deviation (SD). Questionnaire results will be compared against different baseline characteristics of the studied group. According to the type and distribution of data, suitable tests for inferential statistics will be used. Significance of the results will be presented in the form of P-value.

ELIGIBILITY:
Inclusion Criteria:

* hepatologists

Exclusion Criteria:

* Non hepatologists

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hepatologists
Sampling Method: Probability Sample
Enrollment: 717 (Actual)
Dates: Start 2013-08; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Hepatic fibrosis | 3 years
  Percentage of hepatologists accepting invasive versus non-invasive methods for assessment of hepatic fibrosis and cirrhosis.

SECONDARY OUTCOMES:
Trust in non-invasive methods | 3 years
  Percentage of hepatologists trusting invasive versus non-invasive methods for assessment of hepatic fibrosis and cirrhosis.
use of non-invasive methods | 3 years
  Percentage of hepatologists who use invasive versus non-invasive methods for assessment of hepatic fibrosis and cirrhosis.
combining non-invasive methods | 3 years
  Percentage of hepatologists combining different non-invasive methods for assessment of hepatic fibrosis and cirrhosis.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Alboraie, M.Sc, Principal Investigator — Al-Azhar University
Locations (1):
- Al-Azhar Uinversity, Cairo, Cairo Governorate, Egypt